CLINICAL TRIAL: NCT05926804
Title: A Randomized "Screen and Treat" Helicobacter Pylori Eradication Trial in 14-18 Years Old Adolescents Residing in Three Regions of Chile: Effectiveness and Microbiological-host Implications
Brief Title: A "Screen and Treat" Helicobacter Pylori Eradication Trial in Adolescents in Three Regions of Chile
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miguel O'Ryan Gallardo (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor-Investigator, Miguel O'Ryan Gallardo, Medical Doctor, Pediatrician, Infectious Diseases Specialist. Full Professor., University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1220964; 1220964 (Other Grant/Funding Number: Fondecyt Fondo Nacional de Desarrollo Científico y Tecnológico)
Record Dates: First submitted 2023-06-01; First posted 2023-07-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Screen and treat; Pepsinogen; Adolescent
MeSH Terms: interventions — Lansoprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Screening phase: 14-18-year-old students (up to 1000) from three cities will be invited. After obtaining informed consent, eligible participants without exclusion criteria will undergo an H. pylori screening test (Urea Breath Test; UBT). Those negative will exit, except for a subset to be followed as a non-infected controls. Subjects with a positive test will undergo two confirmatory tests 30 days apart to confirm infection persistence. Approximately 20-25% are expected to be positive.
  Intervention phase: those with persistent H. pylori infection will undergo gastroenterological evaluation 1 month before randomization (2:1) to receive antimicrobial treatment or no treatment. Non-infected controls will be followed at matched intervals. If untreated, subjects with persistent infection will be offered the eradication regimen after completing the initial 6-month follow-up with blood and stool samples taken.
Who Masked: Outcomes Assessor
Masking Description: Blinded Gastroenterologist or trained physician who performs the surveillance after eradication treatment. No other parties will be masked in the clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cases (Experimental): 140 children with H. pylori-persistent infection, who will receive eradication therapy
  Interventions: Drug: Lansoprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Metronidazole
- Controls (No Intervention): 70 children with H. pylori-persistent infection, who will not receive eradication therapy
- Non infected Controls (No Intervention): 60 adolescents with no H. pylori infection, they will not receive eradication therapy

INTERVENTIONS:
Drug: Lansoprazole — 14 days of Lansoprazole (30 mg BID) (days 1-14)
  Arms: Cases
Drug: Amoxicillin — 7 days of Amoxicillin (1000 mg BID) (days 1-7)
  Arms: Cases
Drug: Clarithromycin — 7 days of Clarithromycin (500 mg BID) (days 8-14)
  Arms: Cases
Drug: Metronidazole — 7 days of Metronidazole (500 mg BID) (days 8-14)
  Arms: Cases

SUMMARY:
Gastric cancer remains a global health problem, and Chile has one of the highest GC mortality rates in the region. Helicobacter pylori (H. pylori) infection is ubiquitous in Chilean adults, and it constitutes the main cause of GC worldwide. A long-term process occurs from premalignant lesions to carcinoma. H. pylori eradication during early stages of disease significantly impacts outcomes, favoring survival, disease reversal and molecular changes, which supports a "screen and treat" strategy in asymptomatic populations in areas with intermediate-to-high GC prevalence. The Investigators' previous research has shown that H. pylori infection is acquired in early childhood with low rates of spontaneous eradication. A pilot treatment study in a subset of school-aged asymptomatic children showed a high rate of successful eradication (>95%), good tolerance, and was associated with a decrease in serum biomarkers of gastric damage (pepsinogen I and II). Based on the results of these studies, the Investigators propose to advance towards the next stage of this research process: a "screen and treat" strategy. The current trial starts with a Screening phase testing up to 1000 asymptomatic adolescents 14-18 years of age from 3 cities of Chile (Colina, Temuco and Coyhaique), to find a total of 210 persistently-infected participants. Persistently-infected adolescents will be included in a Second phase of this trial: A randomized, case-control, non-blinded study to either receive antimicrobial treatment targeting H. pylori eradication (cases) or no treatment (controls). A subset of 60 non-infected adolescents will be followed-up in matched times. This aims to provide evidence on the effect of treatment on clinical outcomes and serum biomarkers related to gastric damage, as well as composition and antimicrobial resistance of gut microbiota. The Investigators expect that eradication therapy will be successful in >90% of persistently infected adolescents, with reinfection rates not surpassing 15% in a 2-3 year period, and to be associated with a decrease in clinical findings indicative of gastric disease, and a decrease in serum biomarker indicative of "gastric damage".

DETAILED DESCRIPTION:
Background: Helicobacter pylori (H. pylori) infection is the main cause of gastric cancer (GC), and long-term process occurs from premalignant lesions to carcinoma. H. pylori eradication during early stages of disease in young adults ("screen and treat") significantly impacts GC favoring survival, disease reversal and molecular changes. Effects of eradication therapy in affecting gut microbiome diversity and composition, and increasing antibiotic resistance rates in commensal bacteria, appear to be transient in most studies. The investigators have shown that infection is acquired mainly during the first 5 years of life, most infected children remain persistently infected with low rates of spontaneous eradication and persistently infected children have more abdominal complaints and higher levels of pepsinogen (PG) II (marker of gastric damage). A pilot eradication trial in persistently infected school-aged children showed that with sequential triple therapy, eradication was achieved in 96.8% of children, and treated children had a decrease in PG I and II levels compared to non-treated. The Investigators propose a "screen and treat" strategy aimed at a transition age between childhood and adulthood, in areas with intermediate-high gastric cancer prevalence, to assess efficacy of eradication, its clinical and molecular benefits and potential microbial side effects. Aims: The primary aim will be to determine the effectiveness of H. pylori eradication therapy in 14-18 years old adolescents in three regions with nearly 20-25% persistence rates, and determine the effect of eradication on clinical and serum biomarkers of gastric disease/damage. The secondary aims will be to determine the effects of H. pylori eradication therapy on antimicrobial resistance of potentially pathogenic enteric bacteria, and on gut microbiome composition. Exploratory aims: To determine the presence of clarithromycin resistance genes in H. pylori by stool analysis of children not achieving eradication, and determine the effects of reinfection on clinical findings indicative of gastric disease, and biomarkers indicative of "gastric damage", gut microbiota composition and antimicrobial resistance of H. pylori and other potentially pathogenic bacteria. Methods: The Investigators will invite, through contact with the health and educational authorities of Colina, Temuco and Coyhaique, 14-18 year old students until we reach up to 1000 adolescents enrolled. H. pylori screening test (Urea Breath Test; UBT) will be offered, and adolescents with a positive test will undergo two additional tests, separated by 30 days, in order to confirm infection persistence (at least two positive tests). It is expected that 20-25% of adolescents screened to be positive for H. pylori, of which over 90% will be persistently infected. 210 Subjects with persistent infection will then be randomized 2:1 to receive either an antimicrobial course targeting H. pylori eradication (7 days of lansoprazole and amoxicillin followed by 7 days of lansoprazole and clarithromycin plus metronidazole) or no treatment. Participants will be followed-up with UBT (1 month post treatment, and then every 6 months for the remaining surveillance period), gastroenterological evaluation (2 weeks pre treatment, 1 month, 3 months, 9 months and 18 months post treatment), blood samples and stool samples (2 weeks pre-treatment, 1 month and 6 months post treatment). A subset of 60 non-infected students from each site will be followed-up in matched times. To those subjects with persistent infection who do not receive treatment, the same eradication regimen will be offered after they have completed the initial 6-month follow-up with their blood and stool samples taken.

Serum gastric damage biomarkers will be assessed using GastroPanel® (PGI, PGII, Gastrin) and ELISA commercial kits (VCAM-1, CXCL13). Escherichia coli and Enterococcus spp will be cultured from stools samples, and resistance to 6 antimicrobials will be assessed by disk diffusion method. H. pylori clarithromycin resistance gene will be amplified from stools using nested-qPCR. Composition of gut microbiome will be characterized by amplification and sequencing the 16SrRNA gene from stools, ant then bioinformatics analysis. Expected results: The prevalence of persistent H. pylori infection will be around 20-25% in adolescents from Colina, Coyhaique and Temuco. Eradication will be successful in >90% of persistently infected students, and reinfection rates will not surpass 15% in a 2-3 year period. Eradication will be significantly associated with a decrease in clinical findings indicative of gastric disease, and a decrease in biomarker levels indicative of "gastric damage". Treatment will have a transitory effect on increasing antimicrobial resistance rates of potentially pathogen enteric bacteria (Escherichia coli, Enterococcus spp.). Treatment will have a transitory effect on disrupting gut microbiota composition at phylum, class, order, family and genus levels, which will be restored to levels comparable to non-infected healthy teenagers at the end of follow-up. In those adolescents for whom eradication therapy fails, clarithromycin resistance will be more prevalent in pretreatment samples compared to those eradicating H. pylori; in reinfected children, treatment will have a transitory effect on increasing detection rates of H. pylori clarithromycin resistance genes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy teenagers 14-18 years of age from Colina, Temuco or Coyhaique
2. At least one responsible adult family member accessible for phone contact.
3. Persistent H. pylori infection determined by at least 2 positive UBT tests in a 3 months period (except for Non-infected Controls)

Exclusion Criteria:

1. Teenagers not consenting to treatment will be invited to continue as non-treated controls.
2. Known allergy to any of the antimicrobials used in the trial protocol (except for Non-infected Controls)
3. Signs/symptoms compatible with organic abdominal pain according to Rome IV criteria: persistent right upper or right lower quadrant pain, dysphagia, odynophagia, persistent vomiting, gastrointestinal blood loss, involuntary weight loss, deceleration of linear growth, delayed puberty.
4. Prior eradication therapy
5. Antimicrobial course received during the previous month (at least 3 days of treatment at appropriate dosing, children meeting this criteria can be included at a later stage)
6. Pregnancy
7. Use of immunosuppressive or biologic drugs
8. Children deemed "not healthy" after review of the questionnaire by study physician

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of persistently-infected teenagers which change UBT status from positive to negative 1 month post-treatment, as compared to non-treated subjects. | a. Baseline: 2 or 3 samples obtained pre-treatment (separated by 30 days) to detect persistently infected children b. One month post-treatment.
  UBT samples will be obtained pre-treatment and 1 month post-treatment.
Change in the percentage of persistently-infected adolescents which have "gastric disease" according to gastroenterologist examination from baseline (pre-treatment) to 2-4 months post successful eradication therapy, as compared to non-treated subjects | a. Baseline evaluation during the month prior to treatment. b. 2-4 months post treatment
  Clinical evaluation by gastroenterologist or trained physician, blind to the treatment arm of the subject, for specific GI signs/symptoms, will be performed at baseline (during the month prior to treatment) and posttreatment (2-4 months post treatment). Successful eradication: Negative UBT sample 30 days after treatment
Change in blood levels of biomarkers indicative of gastric damage in adolescents with successful eradication after treatment, as compared to non-treated subjects after 6 month follow up. | a. Baseline: Within 2 weeks before initiation of eradication treatment and at similar time-frame in non-treated age matched controls (pre-sample) b. 1 month after treatment c. 6 months post treatment
  Blood samples for Pepsinogen (PG) I, PGII, gastrin and other potential biomarkers of "gastric damage. PGI/PGII/Gastrin-17: will be assessed in serum using GastroPanel® (Biohit Oyj, Helsinki, Finland). Two additional biomarkers of GC will be assessed by ELISA-commercial kits: VCAM-1 and CXCL13. Samples will be collected at baseline, 1 month and 6 months post treatment.

SECONDARY OUTCOMES:
Change in faecal Escherichia coli and Enterococcus antimicrobial resistance rates in treated subjects from baseline to 1 month and 6-12 months post treatment, as compared to non-treated subjects. | a. Baseline: Within one month before treatment b. 1 month post treatment c. 6-12 months post treatment (and at similar time-frame in non-treated age matched controls)]
  Phenotypic antimicrobial susceptibility analysis of Escherichia coli and Enterococcus will be performed from stool samples obtained in both Cases and Controls by Kirby Bauer disc diffusion method. According to patterns of AMR of each bacteria, and the antimicrobials used in this trials, E. coli will be tested against clarithromycin, ampicillin, ampicillin-sulbactam, cefazolin, ceftazidime, levofloxacin, and gentamicin; and Enterococcus will be tested against clarithromycin, ampicillin, ampicillin-sulbactam, penicillin, vancomycin and quinopristin/dalfopristin.
Change in gut microbiome alpha-diversity index in treated subjects from baseline to 1 month and 6-12 months post-treatment, as compared to to non-treated subjects. | a. Baseline: Within one month before treatment b. 1 month post treatment c. 6-12 months post treatment (and at similar time-frame in non-treated age matched controls)]
  For microbiome analysis 30 stool samples from each group (Cases and controls) will be obtained pre and post treatment. Changes in gut microbiota composition in stool samples will be analyzed by sequencing of the 16S rRNA V3 to V4 hypervariable region using Illumina

OTHER OUTCOMES:
Prevalence of H.pylori persistent infection in adolescents in Colina, Temuco and Aysén | 2 or 3 samples obtained pre-treatment (separated by 30 days) to detect persistently infected children
  Persistent infection will be defined by at least 2 positive UBT tests in a 3 month period during the screening phase. Two initial UBT tests will be performed separated by 1 month; a third UBT test will be obtained If there is a discordance in results of the first two tests.
Effect of treatment on frequency of clarithromycin resistance comparing those subject who would not eradicate with non-treated individuals | a. Baseline: Within 1 month before eradication b.Within 6 months after the positive UBT sample indicating non-eradication or reinfection.
  Stool evaluation for presence of Clarithromycin resistance genes will be performed in stool samples obtained before eradication (30 in each group), and after the positive UBT sample indicating non-eradication in conjunction with testing of a similar number of non-treated UBT-positive subjects (20 in each group, including 10 treated and non-eradicated subjects). From DNA isolated from stools, qPCR for ureC will be performed to confirm H. pylori infection, and then qPCR to 23SrRNA gene mutations by Taqman probes will be performed.
Overall reinfection rates in adolescents with successful eradication after treatment | a. One month post treatment to assess successful eradication b. 6 months after treatment c. Every 6 months up to 24 months post treatment
  UBT test performed 1 month after the last day of treatment to confirm eradication, and then 6 months after treatment and subsequently every 6 months to evaluate reinfection up to 24 months post treatment. Reinfection: adolescents in whom H. pylori is successfully eradicated post-treatment, but who then become persistently positive during the remainder of the follow-up period
Change in the percentage of adolescents which have "gastric disease" according to gastroenterologist examination from post eradication to post reinfection. | a. 2-4 months post treatment b. 9-12 months post treatment c. 18-24 months post treatment
  Clinical evaluations by a gastroenterologist or trained physician, blinded to the subject's treatment arm, will be conducted after successful eradication (2-4 months post-treatment), and subsequently at 9-12 months and 18-24 months post-treatment to assess specific GI signs and symptoms and their changes in relation to reinfection during this follow-up period.
Change in blood levels of biomarkers indicative of gastric damage post-reinfection as compared to post-successful eradication. | a. 1 month post treatment b. Within 6 months after the UBT sample indicating reinfection.
  A blood sample will be collected within 6 months after the positive UBT sample indicating reinfection. Biomarkers will be analyzed as described in outcome 3.
Change in gut microbiome alpha-diversity index post-reinfection as compared to post-successful eradication | a. 1 month post treatment b. Within 6 months after the UBT sample indicating reinfection
  A stool sample will be collected within 6 months after the positive UBT sample indicating reinfection. Gut microbiome analysis will be performed according to what is described in outcome 5.
Change in faecal Escherichia coli and Enterococcus antimicrobial resistance rates post-reinfection as compared to post-successful eradication. | a. 1 month post treatment b. Within 6 months after the UBT sample indicating reinfection
  A stool sample will be collected within 6 months after the positive UBT sample indicating reinfection. Antimicrobial resistance will be analyzed as described in outcome 4.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel O'Ryan, MD, Principal Investigator — University of Chile
Locations (3):
- Chile (3):
  - Universidad de Aysén, Coyhaique
  - Universidad de Chile, Santiago
  - Universidad de la Frontera, Temuco

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices), will be shared upon request, as well as the study protocol and questionnaires. Previous authorization of the Human Research Ethics Committee at the Faculty of Medicine, University of Chile will be requested.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 36 months after the publication of results in a peer-reviewed journal
Access Criteria: Data will be shared to researchers who provide a methodologically rigorous proposal and an ethics approval for the project. Proposals should be directed to moryan@uchile.cl, ylucero@uchile.cl, and sgeorge@uchile.cl. To gain access, data requestors will need to sign a data access agreement. Data will be sent via email directly to the person requesting the data.

REFERENCES:
- [Background] O'Ryan ML, Lucero Y, Rabello M, Mamani N, Salinas AM, Pena A, Torres-Torreti JP, Mejias A, Ramilo O, Suarez N, Reynolds HE, Orellana A, Lagomarcino AJ. Persistent and transient Helicobacter pylori infections in early childhood. Clin Infect Dis. 2015 Jul 15;61(2):211-8. doi: 10.1093/cid/civ256. Epub 2015 Apr 2. PMID 25838286
- [Background] O'Ryan ML, Rabello M, Cortes H, Lucero Y, Pena A, Torres JP. Dynamics of Helicobacter pylori detection in stools during the first 5 years of life in Chile, a rapidly developing country. Pediatr Infect Dis J. 2013 Feb;32(2):99-103. doi: 10.1097/INF.0b013e318278b929. PMID 23076385
- [Background] Lucero Y, Lagomarcino AJ, Torres JP, Roessler P, Mamani N, George S, Huerta N, Gonzalez M, O'Ryan M. Helicobacter pylori, clinical, laboratory, and noninvasive biomarkers suggestive of gastric damage in healthy school-aged children: A case-control study. Int J Infect Dis. 2021 Feb;103:423-430. doi: 10.1016/j.ijid.2020.11.202. Epub 2020 Dec 2. PMID 33278617
- [Background] Lucero Y, Lagomarcino AJ, Torres JP, Roessler P, Mamani N, George SA, Huerta N, Gonzalez M, O'Ryan G M. Effect of Helicobacter pylori eradication therapy on clinical and laboratory biomarkers associated with gastric damage in healthy school-aged children: A randomized non-blinded trial. Helicobacter. 2021 Dec;26(6):e12853. doi: 10.1111/hel.12853. Epub 2021 Sep 15. PMID 34528337
- [Derived] George S, Lucero Y, Cabrera C, Zabala Torres B, Fernandez L, Mamani N, Lagomarcino A, Aguilera X, O'Ryan M. Protocol for a randomised 'screen-and-treat' Helicobacter pylori eradication trial in 14-18-years-old adolescents residing in three regions of Chile: effectiveness and microbiological host implications. BMJ Open. 2025 Jan 30;15(1):e084984. doi: 10.1136/bmjopen-2024-084984. PMID 39890135